CLINICAL TRIAL: NCT03192657
Title: Basiliximab as a Treatment of Interstitial Pneumonia in Clinical Amyopathic Dermatomyositis Patients
Brief Title: Basiliximab Treating Interstitial Pneumonia of CADM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADM01
Record Dates: First submitted 2017-06-15; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Lung; Disease, Interstitial, With Fibrosis; Dermatomyositis
MeSH Terms: conditions — Disease; Dermatomyositis | interventions — Basiliximab; Calcineurin Inhibitors; Steroids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basiliximab group (Experimental): 1. Basiliximab: 20mg injection each time at day1 and day5, respectively. The first administration should be within 8 weeks after disease onset.
  2. Calcineurin inhibitors: cyclosporin A 3-5mg/kg/d or tacrolimus 0.05-0.10mg/kg/d.
  3. Steroids: 1mg/kg/d, calculated with prednisone.
  Interventions: Drug: Basiliximab; Drug: Calcineurin Inhibitors; Drug: Steroids
- control group (Active Comparator): 1. Calcineurin inhibitors: cyclosporin A 3-5mg/kg/d or tacrolimus 0.05-0.10mg/kg/d.
  2. Steroids: 1mg/kg/d, calculated with prednisone.
  Interventions: Drug: Calcineurin Inhibitors; Drug: Steroids

INTERVENTIONS:
Drug: Basiliximab — The first administration should be within 8 weeks after disease onset.
  Arms: Basiliximab group
Drug: Calcineurin Inhibitors — Researchers can choose cyclosporin A or tacrolimus according to patient tolerance. Either agent should be applied promptly once infection is ruled out for a patient.
Drug: Steroids — Dosage of steroid can be adjusted according to personal experience of the researcher.

SUMMARY:
This is a 52-week, randomized, open and routine treatment controlled study. This study will assess the safety and efficacy of basiliximab as an add-on treatment for interstitial pneumonia in clinical amyopathic dermatomyositis (CADM) patients. 100 CADM patients are planned to be enrolled in a single center.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill Sontheimer-Bohan-Peter diagnosis criteria for dermatomyositis.
* Agreement of contraception.
* Serum creatine Kinase ≤ 1.5 fold of upper normal level.
* Interstitial pneumonia:

(meet at least two in four of following)

1. interstitial pneumonia images in high resolution CT;
2. DLCO (diffusing capacity)≤ 60% predict in lung function test;
3. elevated serum KL-6;
4. serum anti-MDA5 (+).

Exclusion Criteria:

* Previous application of immunosuppressives or any target treatment for dermatomyositis.
* Clinically significant active infection including ongoing and chronic infections History of human immunodeficiency virus (HIV).
* Confirmed Positive tests for hepatitis B or positive test for hepatitis C Active tuberculosis.
* Abnormal renal function at screening (serum creatine>300μmol/L，or eGFR<60mL/min/1.73m2, or end-stage renal disease).
* Abnormal liver function test at screening (ALT, AST or total bilirubin over 2 fold of upper normal level.
* History of any malignancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Survival | 52 week

SECONDARY OUTCOMES:
Forced vital capacity | 52 week
  measured with lung function test equipment
Total lung capacity | 52 week
  measured with lung function test equipment
Diffusing capacity | 52 week
  transfer factor of the lung for carbon monoxide, measured with lung function test equipment.
Lung CT change | 52 week
  Patient lung high resolution CT images will be semi-quantitatively assessed. Changes over baseline and endpoint will be then calculated.
Serum ferritin | 52 week
Serum KL-6 | 52 week
  A new biomarker of alveolar injury.

CONTACTS AND LOCATIONS:
Locations (1):
- RenJi Hospital, Shanghai, Shanghai Municipality, China